CLINICAL TRIAL: NCT06313801
Title: The Single-center Randomized Study "Comparison of Safety and Effectiveness of the First Line of Polychemotherapy and Polychemotherapy in Combination With PIPAC Sessions in Primary Gastric Cancer With Isolated Peritoneal Carcinomatosis.
Brief Title: Comparing the Safety and Efficacy of First-line Polychemotherapy and Polychemotherapy in Combination With PIPAC Sessions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nizhny Novgorod Regional Clinical Oncology Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPNCD-2309
Record Dates: First submitted 2023-11-15; First posted 2024-03-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer
Keywords: FLOT; mFLOT; dPIPAC; PIPAC
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil; Laparoscopy

STUDY DESIGN:
Intervention Model Description: In the control group, after diagnostic laparoscopy, 6 courses of PCT FLOT are carried out, examination every 3 courses with the performance of control diagnostic laparoscopy after 6 courses of PCT. In the study group, after diagnostic laparoscopy, FLOT PCT courses (1st, 3rd, 5th courses), mFLOT (2nd, 4th, 6th courses) are conducted, examination every 3 courses with dPIPAC sessions with docetaxel (excluding it from systemic administration) on the 2nd, 4th, 6th courses of PCT. In group 2, the function of control laparoscopy is performed by revision at the dPIPAC session of the 6th course of PCT. In both groups, with complete regression of foci along the peritoneum and Cy- in peritoneal lavage - dynamic observation or cytoreductive surgery, with incomplete response - dynamic observation before progression, with progression - the 2nd line of CT or optimal palliative care options.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): FLOT: Docetaxel 50 mg/m2 intravenously on day 1 + Oxaliplatin 85 mg/m2 intravenously on day 1 + Calcium folinate 200 mg/m2 2-hour intravenous infusion on day 1 + fluorouracil 2600 mg/m2 x intravenous infusion 24-hours (infusion of the same of the total dose of fluorouracil for 48 hours) on day 1. Repeat every 2 weeks. 6 courses.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Calcium folinate; Drug: Fluorouracil; Procedure: Diagnostic laparoscopy
- Study group (Experimental): mFLOT: Oxaliplatin 85 mg/m2 intravenously on day 1 + Calcium folinate 200 mg/m2 2-hour intravenous infusion on day 1 + fluorouracil 2600 mg/m2 x intravenous infusion 24-hours (infusion of the same of the total dose of fluorouracil for 48 hours) on day 1. Repeat every 2 weeks. 6 courses.
  + The drugs for PIPAC - Docetaxel 50 mg/ m2 diluted with saline sodium chloride to a total volume of 200 ml (intraperitoneal pressurized infusion).
  Interventions: Drug: Oxaliplatin; Drug: Calcium folinate; Drug: Fluorouracil; Procedure: Diagnostic laparoscopy; Combination Product: dPIPAC ( The description of the standard diagnostic laparoscopy procedure and the session of PIPAC (dPIPAC)).

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50 mg/m2 intravenously on day 1
  Arms: Control group
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 on Day 1
Drug: Calcium folinate — 200 mg/m2 2-hour intravenous infusion on day 1
Drug: Fluorouracil — 2600 mg/m2 x intravenous infusion 24-hours (infusion of the samee of the total dose of fluorouracil for 48 hours) on day 1.
Procedure: Diagnostic laparoscopy — Access to the abdominal cavity by Hassen (3 trocars). Carboxyperitoneum - 12 mm of water column - stable pressure maintenance throughout the operation. Revision. Photo recording of 4 quadrants of the abdominal cavity from the paraumbilical port. The evaluation of the PCI index. The evaluation of other distant dissemination. Standard peritoneal lavage of 300 ml Sol. NaCl 0.9 % (37 ºС), with the exposure of 3-5 minutes (with Trendelenburg and Fowler position alternately) and the lavage aspiration, the transfer of the lavage for the cytological examination. Biopsy of perioneal lessions if needed.The operation is completed as standard with the extraction of laparoports and suturing of laparoport wounds.
Combination Product: dPIPAC ( The description of the standard diagnostic laparoscopy procedure and the session of PIPAC (dPIPAC)). — Diagnostic laparoscopy described earlier and PIPAC session. The drugs for PIPAC - Docetaxel 50 mg/ m2 diluted with saline sodium chloride to a total volume of 200 ml. The rate of administration is 30 ml per minute. The maximum pressure in the injector system is 250 PSI. After the spray stage, the exposure is 30 minutes while maintaining the declared intraperitoneal pressure. After the exposure stage, only gas is removed from the abdominal cavity. The operation is completed as standard with the extraction of laparoports and suturing of laparoport wounds.
  Arms: Study group

SUMMARY:
After the initial diagnostic laparoscopy the Control group patients undergo 6 courses of polychemotherapy according to the FLOT scheme; the examination is carried out every 3 courses (after the 3rd and the 6th courses) with the control diagnostic laparoscopy after 6 courses of polychemotherapy. In the event of the complete regression of foci along the peritoneum and receiving Cy- in the peritoneal lavage, the dynamic observation or cytoreductive surgery is considered (optionally); in case of the incomplete response the dynamic observation is carried out until progression; in case of progression the 2nd line of chemotherapy or the optimal palliative care options depending on the clinical situation is considered.

After the initial diagnostic laparoscopy the Study group patients undergo courses of polychemotherapy according to the scheme FLOT (the 1st, the 3rd, the 5th courses) and mFLOT (the 2nd , the 4th, the 6th courses) in the amount of 6 (six, 3+3); the examination is carried out every 3 courses (after the 3rd and the 6th courses) with dPIPAC sessions using docetaxel (thus excluding it from the system administration) in the 2nd , the 4th, the 6th courses of polychemotherapy. Control diagnostic laparoscopy is not performed in the group No 2, its function is performed by the revision at the PIPAC session of the 6th course of polychemotherapy, which corresponds to the time interval of the Control group. In the event of the complete regression of foci along the peritoneum and receiving Cy- in the peritoneal lavage, the dynamic observation or cytoreductive surgery is considered (optionally); in case of the incomplete response the dynamic observation is carried out until progression; in case of progression the 2nd line of chemotherapy or the optimal palliative care options depending on the clinical situation is considered.

DETAILED DESCRIPTION:
Signing the informed consent to participate in the study. All the patients with suspected peritoneal carcinomatosis (according to the results of radiation diagnostics, as well as confirmed peritoneal carcinomatosis by puncture biopsy or by taking ascitic fluid) undergo diagnostic laparoscopy at the first stage. In addition, screening will include all the patients with locally advanced gastric cancer undergoing laparoscopy prior to planning combination treatment. If they have foci of carcinomatosis in the peritoneum PCI up to 15 inclusive and/or Cy+ (as the only manifestation of M1), the patients of this group can be included in the study. The methodology for performing diagnostic laparoscopy is described below (excluding dPIPAC components). Note - the examination of the omental bursa as part of diagnostic laparoscopy is optional, depending on the clinical situation. Screening and examination of patients according to current clinical guidelines for nosology stomach cancer taking into account the examination criteria specified in this protocol. Performing initial diagnostic laparoscopy at the stationary stage according to the standard procedure (described above). If carcinomatosis is detected the evaluation of PCI is carried out by Sugarbaker. The patient randomization based on positive (Cy+) abdominal flushing and/or peritoneal dissemination with PCI index <16. The randomization will be carried out using an Internet resource https://www.sealedenvelope.com. Taking into account the planned set and heterogeneity of the groups, the patients will be stratified before randomization according to the following factors: microscopic carcinomatosis of Cy+ only, macroscopic carcinomatosis PCI up to 7 inclusive, macroscopic carcinomatosis PCI from 8 to 15 inclusive; accordingly, the patients within the strata will be randomized separately.

The Control group (the group No 1). Within 1-4 weeks after the initial diagnostic laparoscopy the group No 1 patients start polychemotherapy courses according to the FLOT scheme in the amount of 6 (six); the examination is carried out every 3 courses (after the 3rd and the 6th courses) with the control diagnostic laparoscopy after 6 courses of polychemotherapy for no more than 2 weeks with no obvious signs of progression (in this case, the patient switches to the 2nd line of chemotherapy). The evaluation of the therapeutic pathomorphosis of foci in the peritoneum is carried out according to the PRGS system (Peritoneal Regression Grading Score). As the result of the treatment: in the event of the complete regression of foci along the peritoneum and receiving Cy- in the peritoneal lavage, after the completion of the planned treatment, the patients switch to the dynamic observation or cytoreductive surgery is considered within 1 month after the completion of polychemotherapy (optionally, by decision of the local council); in case of the incomplete response (due to the immeasurable characteristics of the tumor and the impossibility of evaluation by RECIST), the dynamic observation is carried out until progression; in case of progression the 2nd line of chemotherapy (the scheme at the discretion of the attending physician) or the optimal palliative care options depending on the clinical situation is considered; accordingly the patient completes the therapy proposed by the study. The response criteria are specified separately. Shifting the timing of chemotherapy up to 10 days and the timing of control examinations up to 10 days due to objective circumstances is considered acceptable within the study.

The Study group (the group No 2). Within 1-4 weeks after the initial diagnostic laparoscopy the group No 2 patients start polychemotherapy courses according to the scheme FLOT (the 1st , the 3rd, the 5th courses) and mFLOT (the 2nd, the 4th, the 6th courses) in the amount of 6 (six, 3+3); the examination is carried out every 3 courses (after the 3rd and the 6th courses) with with dPIPAC sessions using docetaxel the examination is carried out every 3 courses (after the 3rd and 6th) with the performance of dPIPAC sessions using docetaxel (thus excluding it from the system administration) in the 2nd , the 4th, the 6th courses of polychemotherapy (all the procedures are performed according to the method described in the protocol; the evaluation of the therapeutic pathomorphosis of lesions in the peritoneum is carried out according to the PRGS system (Peritoneal Regression Grading Score)). Control diagnostic laparoscopy is not performed in the group No 2, its function is performed by the revision at the PIPAC session of the 6th course of polychemotherapy, which corresponds to the time interval of the group No 1. As the result of the treatment: in the event of the complete regression of foci along the peritoneum and receiving Cy- in the peritoneal lavage, after the completion of the planned treatment, the patients switch to the dynamic observation or cytoreductive surgery is considered after the completion of polychemotherapy (optionally, by decision of the local council); in case of the incomplete response (due to the immeasurable characteristics of the tumor and the impossibility of evaluation by RECIST), the dynamic observation is carried out until progression; in case of progression the 2nd line of chemotherapy (the scheme at the discretion of the attending physician) or the optimal palliative care options depending on the clinical situation is considered; accordingly the patient completes the therapy proposed by the study. The method of performing the surgical manual is specified separately. The response criteria are specified separately. Shifting the timing of chemotherapy with dPIPAC sessions up to 10 days and the timing of control examinations up to 10 days due to objective circumstances is considered acceptable within the study.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of signed informed voluntary consent of the patient
2. Age ≥18 years and ≤75 years
3. ECOG ≤1
4. Histological verification of gastric cancer and esophageal-gastric junction Siewert III (adenocarcinoma, ring-cell carcinoma)
5. Her2-neu negative tumor status
6. The presence of a preserved informative block of the primary tumor in the histological archive of the NOCOD (performing a biopsy and/or providing archival material - with the consent of the patient)
7. Verified gastric cancer (adenocarcinoma, ring-cell carcinoma) with the presence of M1 (with the only manifestation of M1 in the form of - Cy+ in initial peritoneal lavage and/or peritoneal dissemination PCI <16)
8. Peritoneal adhesion index PAI <16
9. Absence of active infectious, mental diseases, pronounced allergic conditions, as well as other concomitant pathology that may interfere with the implementation of the therapeutic and diagnostic measures provided for in the protocol
10. Adequate organ function (evaluation by laboratory parameters at screening - evaluation of hemoglobin, neutrophils, platelets, AST, ALT, total bilirubin, urea, creatinine)
11. Consent of men and women with preserved childbearing potential to use highly effective methods of contraception.

Exclusion Criteria:

1. Lack of informed voluntary consent of the patient
2. Age <18 years and >75 years
3. ECOG ≥2
4. Histological forms other than adenocarcinoma and ring-cell carcinoma of the stomach and esophageal-gastric junction Siewert III
5. Her2-neu positive tumor status
6. The absence of a preserved informative block of the primary tumor in the histological archive of the NOCOD
7. M1 with the exception of Cy+ in initial peritoneal lavage and/or peritoneal dissemination PCI <16 (Distant metastases, including mts in supraclavicular, mediastinal, paraaortic (16 collector), ovarian metastases. Note - MTS in peripheral lymph nodes require a fine needle puncture with cytological examination for verification. In case of mts lesions of intracorporeal lymph nodes, the criteria of mts will be - dimensions of more than 15 mm along the short axis or mts-altered structure of the lymph node, regardless of size; PCI ≥16)
8. Peritoneal adhesion index PAI ≥16
9. Contraindications to performing diagnostic laparoscopy
10. Complicated primary tumor (bleeding, decompensated stenosis, dysphagia III-IV) if not corrected.
11. Decompensated concomitant pathology
12. Primary multiple tumors (except basal cell skin cancer and cervical cancer in situ - provided there are no signs of relapse of the disease)
13. Any specific antitumor treatment for stomach cancer and /or other malignant tumor in the anamnesis (except basal cell skin cancer and cervical cancer in situ - provided there are no signs of relapse of the disease)
14. Previous specialized treatment for stomach cancer
15. Known individual intolerance to drugs included in the protocol
16. Pregnancy, breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival. | 4 years 6 months
  Time interval from randomization to progression of disease, death from any cause or date of last observation in the absence of these events. In months with an accuracy of 0.1. (Time Frame: 4 years 6 months)
Complications from polychemotherapy. | 3 years 6 months
  Complications from polychemotherapy (including intraperitoneal administration), evaluated according to СТСАЕ v5.0. The proportion of patients with any adverse events; the proportion of patients with grade 3-5 adverse events; the proportion of patients with complications in qualitative terms (for example: hematological, gastrointestinal, etc.). (Time Frame: 3 years 6 months)

SECONDARY OUTCOMES:
The overall survival. | 4 years 6 months
  Time interval from randomization to death from any cause or date of last observation in the absence of these events. In months with an accuracy of 0.1. (Time Frame: 4 years 6 months)
The completeness of the planned therapy. | 3 years 6 months
  The proportion of patients who received all the therapy planned in the study in each group. (Time Frame: 3 years 6 months)
Percentage of patient conversions to Су- and PCI- rate. | 3 years 6 months
  The proportion of patients conversions to Су- and PCI- rate (Time Frame: 3 years 6 months)
Surgical complications of operated patients | 3 years 6 months
  Surgical complications of operated patients (the evaluation by Clavien-Dindo classification) (the proportion of patients with surgical complications IIIb-V grade). (Time Frame: 3 years 6 months)
Аssessment of the quality of life | 4 years
  Quality of life assessment by European Organisation for Research and Treatment of Cancer scale (unabbreviated scale title) Quality of Life Questionnaire - Core 30 (QLQ-C30) by Scoring of the QLQ-C30 Summary Score using the descriptive analysis with the qlqc30 command (detailed description in manual ISBN 2-9300 64-22-6). The minimum values of general health score are mean a worse outcome (minimum score 0), the maximum values of general health score are mean a better outcome (maximum score 100). (Time Frame: 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Gamayunov, DMS, Study Director — Chief oncology specialist in the region
Locations (1):
- Research Institute of Clinical Oncology "Nizhny Novgorod Regional Clinical Oncological Dispensary", 11/1, Delovaya street, Nizhny Novgorod, 603126, Nizhny Novgorod, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT06313801/Prot_SAP_000.pdf